CLINICAL TRIAL: NCT05579015
Title: Predicting Illness Trajectories In Fully Remitted Major Depression Using Concurrent TBS/fNIRS
Acronym: TBS/fNIRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSEARS20220812002
Record Dates: First submitted 2022-09-14; First posted 2022-10-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Major Depression in Remission; Healthy
Keywords: Theta-burst stimulation; Remitted depression; Relapse prediction; Functional NIRS; Concurrent TBS/fNIRS
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rMDD group (Experimental): Participants with remitted MDD who will receive concurrent TBS/fNIRS with iTBS and followed by cTBS after one hour. This group will also receive follow-up telephone interviews every 3 months for 2 years to monitor major depressive episode recurrence.
  Interventions: Device: Theta-burst stimulation (TBS); Other: telephone interviews
- Healthy control group (Other): Healthy participants who will receive TBS/fNIRS with iTBS and followed by cTBS after one hour. No follow-up interviews will be conducted for this group.
  Interventions: Device: Theta-burst stimulation (TBS)

INTERVENTIONS:
Device: Theta-burst stimulation (TBS) — TBS comprises 3-pulse 50-Hz bursts, applied every 200 ms (at 5 Hz), as described previously. iTBS consists of 2-second trains with an inter-train interval of 8 seconds. The investigators will repeat the trains (30 pulses; 10 bursts) 20 times to reach a total number of 600 pulses (3x10x20). cTBS will comprise uninterrupted bursts to reach a total of 600 pulses. Concurrent TBS/fNIRS stimulation will be applied over the left (iTBS) and right (cTBS) DLPFC at an intensity of 90% resting motor threshold (RMT). This corresponds to ~110% of the active motor threshold. Stimulation at 90% RMT will also ensure compliance, reduce sensory discomfort and minimize dropout rates. Still, scalp discomfort will be recorded directly after the stimulation. The stimulation site over the DLPFC will be determined using the international 10-20 system and correspond to the F3 label.
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)
Other: telephone interviews — Telephone interviews will be conducted at the follow-up stage. RMDD group will receive follow-up telephone interviews every 3 months for 2 years to monitor major depressive episode recurrence
  Arms: rMDD group

SUMMARY:
Major depressive disorder (MDD) is the world's leading cause of disability according to the World Health Organization. MDD is highly recurrent, even if clinical remission is reached after successful treatment. In fact, the enormous burden of disability, mortality and financial costs is due to the recurrent and chronic nature of MDD. The reliable prediction of the recurrence of major depressive episodes (MDEs) based on a prognostic model that is informed by biological, neurophysiological or neuroimaging data would be valuable and lifesaving for many. However, such models are still lacking.

Several lines of evidence point to abnormal prefrontal control over limbic emotion processing areas in MDD owing to diminished prefrontal excitability that seems to persist during MDD remission (rMDD). Prefrontal excitability in rMDD may thus be a trait marker of MDD and may potentially be indicative of disease recurrence. Yet, research investigating the potential utility of prefrontal excitability for predicting the recurrence of MDEs is lacking. Cortical excitability can be investigated using transcranial magnetic stimulation (TMS); however, human studies have mostly probed cortical excitability of the motor cortex, a brain region not considered to be central in the neuropathology of MDD. Hence, knowledge of the effect of TMS on prefrontal excitability is limited. Moreover, whether immediate prefrontal modulation by TMS can predict the recurrence of MDEs in fully remitted MDD patients remains to be investigated. Thus, there is a need for research that aims to quantify the direct and immediate aftereffects of TMS on prefrontal function. Most importantly, with regard to precision medicine, there is a need for research that explores the utility of immediate prefrontal reactivity to TMS for predicting MDE recurrence. Here, the investigators propose a research program that will exploit the combination of functional near-infrared spectroscopy (fNIRS) with brain stimulation. Concurrent theta-burst stimulation (TBS)/fNIRS measurements will allow us to systematically investigate stimulation-induced modulation of blood oxygenation as a proxy for induced brain activity changes (TBS is a modern form of patterned TMS). The findings from this study will (1) elucidate the immediate effects of excitatory and inhibitory brain stimulation on prefrontal activity in rMDD and controls and (2) validate the potential utility of stimulation-induced brain modulation for the prediction of MDE recurrence.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of recurrent depressive disorder by an experienced psychiatrist but currently in full remission (ICD 11, 6A71.7) according to results of the Mini International Neuropsychiatric Interview (MINI) and the Patient Health Questionnaire (PHQ-9), with a score ≤ 4;
* at least two previous MDEs within the last 10 years;
* no or stable (≥4 weeks) psychopharmacological medication.

Exclusion Criteria:

* severe internal diseases;
* neurological disorders or a history of severe head injuries;
* current psychiatric comorbidities, including addiction;
* pregnancy;
* common fNIRS and TMS exclusion criteria, such as a history of brain surgery, head injury, cardiac pacemaker, deep brain stimulation, intracranial metallic particles, history of seizures, and antiepileptics and benzodiazepines corresponding to a dose of >1 mg lorazepam/d. Potential participants taking antidepressants will be included if there has been no recent change to either dosage or medication (within 4 weeks).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of a major depressive episode | Up to 2 years.
  Primary clinical outcome measure: recurrence of a major depressive episode (based on MINI and PhQ-9 ≥ 5).
Oxyhemoglobin (HbO) change compared to baseline | During and within 3 minutes post TBS-fNIRS measurement.
  Primary imaging outcome measure: TBS-induced HbO change in the dorsolateral prefrontal cortex (DLPFC) during and after stimulation.

SECONDARY OUTCOMES:
Hemoglobin (Hb) change compared to baseline | During and within 3 minutes post TBS-fNIRS measurement
  Secondary Imaging Outcome Measure: TBS-induced Hemoglobin (Hb) change in the dorsolateral prefrontal cortex (DLPFC) during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Georg S. Kranz, PhD, Principal Investigator — The Kong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request